CLINICAL TRIAL: NCT03690128
Title: Individual Early Warning Score (I-EWS) - Does Clinical Assessment Improve Detection of Acute Deterioration in Hospitalized Patients - a Cluster-randomized Trial
Brief Title: Individual Early Warning Score (I-EWS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Principal Investigator, Associate Professor, Consultant, DMSci, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17017332
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Early Warning Score; Risk Stratification
Keywords: Clinical deterioration; Risk stratification; Patient Safety; Early Warning Score; Monitoring; Clinical assessment
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Intervention Model Description: A prospective, cluster randomized, cross-over, non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm - standard EWS procedure (Active Comparator): Standard use of the current implement Early Warning System, based on the principles of the National Early Warning Score and with a standard escalation protocol.
  Interventions: Behavioral: Standard EWS - Control (Trigger Tool)
- Intervention Arm - I-EWS (Active Comparator): Implementation of Individual Early Warning Score (I-EWS) with a systematic clinical assessment with a standard escalation protocol as intervention 7 parameters (Respiration rate, pulse, saturation, systolic blood pressure, consciousness, temperature, Oxygen) are registered , an aggregated score is generated. In the electronic patient journal (Sundhedsplatformen), the nursing staff is asked to reevaluate the aggregated score based on their clinical assessment of the patient. The aggregated score can be upgraded with up to 6 points and downgraded with up to 4.
  This new I-EWS score interacts with the standard escalation protocol which defines the observation frequency and relevant clinical actions.
  Interventions: Behavioral: I-EWS with incorporated clinical assessment (Trigger Tool)

INTERVENTIONS:
Behavioral: I-EWS with incorporated clinical assessment (Trigger Tool) — In relation to systematic measurement of vital parameters the nursing staff will perform an individual clinical assessment of the patient and adjust the I-EWS score accordingly.
  Arms: Intervention Arm - I-EWS
Behavioral: Standard EWS - Control (Trigger Tool) — Standard EWS - Based on principles of National Early Warning Score (NEWS)
  Arms: Control Arm - standard EWS procedure

SUMMARY:
Early Warning Score (EWS) is a clinical scoring system used in hospitals in Denmark and internationally to systematically observe admitted patients using a standardised response algorithm. Consisting of a score based on the patients' vital signs, it only leaves limited space for individual assessment. Patient safety but also resource utilisation is a key issue in health systems today. We have developed a new individual EWS system (I-EWS) that reintroduces the individual clinical assessment for a more personalised observation. Our hypothesis is that I-EWS will not increase the mortality among hospitalised patients compared to EWS but will improve workflow by reducing unnecessary observations and freeing staff resources, potentially leading to improved patient care. The impact of I-EWS on mortality, the occurrence of critical illness, and usage of staff resources will be evaluated in a prospective, cluster randomised, non-inferiority study conducted at eight hospitals in Denmark.

DETAILED DESCRIPTION:
Every year more than 250,000 patients are admitted in the Capital Region of Denmark. During admissions, the clinical track and trigger system "Early Warning Score" (EWS) is used to systematically observe and detect acutely deteriorating patients. The system is designed to prevent serious adverse events like unanticipated transfer to the intensive care unit, cardiac arrest and unexpected death. EWS consists of standardized measurements of the patient's vital signs and an escalation protocol that determines further actions based on the aggregated EWS score. At admission, and as a minimum twice a day, nurses measure vital signs on all hospitalized patients. Depending on the predetermined cut-off values (i.e. heart rate above 150 bpm = 3 points) an aggregated score is calculated. Based on the total score, the escalation protocol determines the time interval for the next measurement as well as a clinical action (i.e. call for attending doctor). EWS is developed to detect and to treat potentially deterioration of disease that might lead to critical illness and death. In its current form, there is only limited room for individual clinical assessment.

A standardized track and trigger system like EWS does not differentiate between different types of disease or the patient's individual physiological response. Therefore, there is a potential risk that the system fails to detect a patient with an abnormal stress response. Additionally; patients suffering from chronic illness might have different normal values than healthy patients, leading to unnecessarily excess observation, measurement, and suboptimal usage of limited staff resources.

Previous studies have shown that Early Warning System scores perform well for prediction of cardiac arrest and death within 48 hours, although the impact on health outcomes and resource utilization remains uncertain, often owing to methological limitations.

It is possible, but never studied before, whether the combination of vital signs with individual clinical assessment is a better tool for identifying hospitalized high-risk patients than the existing algorithms.

Further improvement and optimizing of the EWS is necessary, as there is potential to improve patient care and use staff resources more appropriate.

The purpose of the study is to investigate the impact of the I-EWS that has a systematic involvement of clinical assessment and the possibility to adjust the score, whilst keeping the same escalation protocol. I-EWS will be compared to the existing EWS with a focus on mortality, critical illness, and the use of staff resources.

Our hypothesis is that I-EWS, where clinical assessment is given a more prominent role will not increase the mortality among hospitalized patients but can reallocate personnel resources.

I-EWS is built in to electronic patient journal system "Sundhedsplatformen" it is only available in Sundhedsplatformen (SP) at hospitals assigned to I-EWS. Four hospitals are randomized to use I-EWS for 6,5 months, the remaining four hospitals are control hospitals using the current EWS in this period.

After 6,5 months a single cross-over will be preformed, and the previous control hospitals will use I-EWS over the next 6,5 months and the previous intervention hospitals, will go back to the current EWS for this period.

EWS scores and subsequent actions are documented in real time in SP. The first two weeks and final four weeks of each period will be excluded due to a implementation period. Data regarding patients, interventions and serious adverse events during hospitalization (i.e., cardiac arrest, the request of MET or unexpected death) will be accessed through SP and the Danish Central Registries (The Danish National Patient Registry, the Civil Registration System, DanArrest). After extraction, all data will be depersonalization and stored at a secured network in accordance with the current guidelines for data management in the Capital Region of Denmark.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥18 years of age admitted more than 24 hours to a ward at participating hospitals will be included.

Participating hospitals are

* Herlev & Gentofte Hospital
* Nordsjaellands Hospital
* Bispebjerg Hospital
* Rigshospitalet, Glostrup - Medical Ward
* Amager & Hvidovre Hospital
* Zealand University Hospital
* Slagelse Hospital
* Holbaek Hospital

Exclusion Criteria:

* Wards not using standard EWS, paediatric, obstetric and intensive, due to they use special variations (Pediatric early warning score, Obstetric Early warning Score or continous monitoring).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150000 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
All Cause mortality at 30 days | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day | Assessed after one year, after completion of the study

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Calculated as days from date of index admission to date of discharge
All Cause mortality at 2 days | 2 days (48 hours) after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All Cause mortality at 7 days | 7 days (168 hours) after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.

OTHER OUTCOMES:
Frequency of changes in I-EWS scores that lead to an escalation or de-escalation in the escalation protocol | Assessed after one year, after completion of the study
Comparison of changes in EWS score due to I-EWS modification (intervention group) and due to temporary or chronic acceptable values (control group) | Assessed after one year, after completion of the study
The number of Cardiac arrests* during hospital stay, reported in numbers (%) | Assessed after one year, after completion of the study
  *Definition - Presence of a clinical cardiac arrest (as defined in the resuscitation guidelines) in patients without a DNAR (Do Not Attempt Resuscitation) order. Registered in DANARREST.
The number of Cardiac arrests* during hospital stay, reported in number per 10,000 ward days | Assessed after one year, after completion of the study
  *Definition - Presence of a clinical cardiac arrest (as defined in the resuscitation guidelines) in patients without a DNAR (Do Not Attempt Resuscitation) order. Registered in DANARREST.
Scores generating a call for Mobile Emergency team (MET) reported in absolute number (%) | Assessed after one year, after completion of the study
Scores generating a call for Mobile Emergency team (MET) reported in absolute per 10,000 ward days | Assessed after one year, after completion of the study
Scores generating a call for the attending doctor, reported in absolute number (%) | Assessed after one year, after completion of the study
Scores generating a call for the attending doctor, reported per 10,000 ward days | Assessed after one year, after completion of the study
All cause mortality - Subgroup analysis of patients admitted to Herlev-Gentofte Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Nordsjaellands Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Bispebjerg Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Glostrup Hospital (Medical Ward) | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Amager-Hvidovre Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Zealand University Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Slagelse Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients admitted to Holbaek Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients Age ≤ 39 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients Age 40 to 69 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients Age ≥ 70 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with cardiovascular disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with cancer disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with pulmonary disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with infectious disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with neurological disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
All cause mortality - Subgroup analysis of patients diagnosed with surgical condition | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Herlev-Gentofte Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Nordsjaellands Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Bispebjerg Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Amager-Hvidovre Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Zealand University Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Slagelse Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients admitted to Holbaek Hospital | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients Age ≤ 39 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients Age 40 to 69 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients Age ≥ 70 years | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with cancer | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with cardiovascular disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with pulmonary disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with infectious disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with neurological disease | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.
The number of NEWS/I-EWS scores per patient per day - Subgroup analysis of patients diagnosed with surgical condition | 30 days after index admission
  Time frame starts at the beginning of the index admission, defined as first admission in the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Iversen, MD, DMSci, Study Director — Department of Cardiology, Herlev Hospital
Locations (8):
- Denmark (8):
  - Bispebjerg Hospital, Copenhagen, Capital Region of Denmark
  - Amager & Hvidovre Hospital, Copenhagen, Capital Region of Denmark
  - Herlev & Gentofte Hospital, Copenhagen, Capital Region of Denmark
  - Rigshospital, Glostrup, Medical Ward, Glostrup Municipality, Capital Region of Denmark
  - Nordsjaellands Hospital, Hillerød, Capital Region of Denmark
  - Holbaek Hospital, Holbæk, Region of Zealand
  - Zealand University Hospital (Roskilde & Køge), Roskilde, Region of Zealand
  - Slagelse Sygehus, Slagelse, Region of Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nielsen PB, Langkjaer CS, Schultz M, Kodal AM, Pedersen NE, Petersen JA, Lange T, Arvig MD, Meyhoff CS, Bestle MH, Holge-Hazelton B, Bunkenborg G, Lippert A, Andersen O, Rasmussen LS, Iversen KK. Clinical assessment as a part of an early warning score-a Danish cluster-randomised, multicentre study of an individual early warning score. Lancet Digit Health. 2022 Jul;4(7):e497-e506. doi: 10.1016/S2589-7500(22)00067-X. Epub 2022 May 19. PMID 35599143
- [Derived] Nielsen PB, Schultz M, Langkjaer CS, Kodal AM, Pedersen NE, Petersen JA, Lange T, Arvig MD, Meyhoff CS, Bestle M, Holge-Hazelton B, Bunkenborg G, Lippert A, Andersen O, Rasmussen LS, Iversen KK. Adjusting Early Warning Score by clinical assessment: a study protocol for a Danish cluster-randomised, multicentre study of an Individual Early Warning Score (I-EWS). BMJ Open. 2020 Jan 7;10(1):e033676. doi: 10.1136/bmjopen-2019-033676. PMID 31915173

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT03690128/SAP_002.pdf